CLINICAL TRIAL: NCT01250860
Title: Short-term Effects of the Simultaneous Use of Two Physiotherapeutic Methods in the Treatment of Adolescent Idiopathic Scoliosis - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Medical University of Silesia, Department of rehabilitation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BW-08-AM
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: The Spirometry;; The Strength of Respiratory Muscles - MIP, MEP;; Kyphosis (Plurimeter-V); The Angle of Trunk Rotation in Thoracic Part
Keywords: Manual therapy; DoboMed exercise; Spirometric test
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Sham Comparator): Control DoboMed group - only specific active exercises: symmetrical positions for exercising; asymmetrical active movements; thoracic spine kyphotization; transverse plane derotation; apical area involvement; concave ribs mobilization; exteroceptive facilitation; respiration-directed movements of the thorax and spine; three-dimensional displacement of vertebra; active autocorrection.
  Interventions: Behavioral: Sham therapy
- Experimental group (Experimental): Experimental DoboMed and Kaltenborn manual therapy. Suitable techniques were chosen according to manual examination: cervical spine; thoracic spine; lumbar spine; costovertebral articles; pelvis position. During the 15 sessions in group "DK" we used:derotational manual terapy techniques in selected segments of spine in preparation for the exercises according to the DoboMed method; the manual techniques used in continuation study were different from techniques in pilot study.
  Interventions: Other: Derotational manual therapy techniques in selected segments in spine

INTERVENTIONS:
Other: Derotational manual therapy techniques in selected segments in spine — Derotational manual therapy techniques in selected segments of spine in preparation for the exercises according to the DoboMed method.
  Arms: Experimental group
Behavioral: Sham therapy
  Arms: Control Group

SUMMARY:
The assessment of influence joint physiotherapy (DoboMed and OMT Kaltenborn - Evjenth) on the function of the respiratory system and the morphology of the ribcage in short-term intensive physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* girls aged 10 to 16
* one arc right side curve
* Cobb range 12 - 40 degrees

Exclusion Criteria:

* bigger Cobb range
* double arc curve
* no parent approval
* lack of cooperation

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Simultaneous use of two physiotherapeutic methods in the treatment of Adolescent Idiopathic Scoliosis | 3 weeks
  Forty-two girls with thoracic AIS; mean age - 14.5y. Cobb - (range 12-40) The group was divided into two randomized subgroups. DoboMed was applied in group "D" only. DoboMed and manual therapy (Kaltenborn) were applied in group "DK". The spirometry, the strength of respiratory muscles (maximal inspiratory and expiratory pressures- MIP, MEP), kyphosis (plurimeter-V) and the angle of trunk rotation (ATR) in thoracic part (Bunnell scoliometer) were estimated twice - before and after therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Silesia, Katowice, Silesian Voivodeship, Poland